CLINICAL TRIAL: NCT07013318
Title: Pre- and Post-Treatment Investigation of B12 and Folic Acid (Folate) Levels in Patients Receiving Antiepileptic (Anticonvulsant) Treatment for Neuropathic Pain: Retrospective Study
Brief Title: Pre- and Post-Treatment Investigation of B12 and Folic Acid (Folate) Levels in Patients Receiving Antiepileptic (Anticonvulsant) Treatment for Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 85
Record Dates: First submitted 2025-05-21; First posted 2025-06-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-05

CONDITIONS: Neuropathic Pain; Vitamin B 12 Deficiency
Keywords: antiepileptic drug; folic acid
MeSH Terms: conditions — Neuralgia; Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuropathic pain (NeP) is a disorder of the nervous system resulting from altered mechanisms operating at the peripheral nervous system, spinal cord and supraspinal levels and is defined by the International Association for the Study of Pain as pain resulting from nervous system pathologies that cause changes in the function, chemistry and structure of neurons . NeP affects 2-8% of the world population and can have a significant impact on the patient's functional abilities and quality of life. NeP can be caused by spinal cord injury, brain and spinal cord tumours and other diseases affecting the nervous system. NeP can be secondary to extremely common conditions such as diabetes, stroke, cancer, herpes zoster virus infection and autoimmune disease. These recommendations were finalised in 2019 and published in April 2020. Following the GRADE system, the recommendations suggest first-line treatment options including serotonin-noradrenaline reuptake inhibitors (duloxetine and venlafaxine), gabapentin, tricyclic antidepressants, and the specialised use of topical lidocaine and transcutaneous electrical nerve stimulation for peripheral neuropathic pain. Pregabalin, tramadol and combination therapy (combining antidepressants with gabapentinoids) are recommended as second-line treatments. Highly concentrated capsaicin patches and botulinum toxin A are recommended as second-line treatments, especially for focal peripheral neuropathic pain. Third-line treatment options include high-frequency repetitive transcranial magnetic stimulation (rTMS) of the primary motor cortex (motor cotex-1/M1), spinal cord stimulation (for failed back surgery syndrome and painful diabetic polyneuropathy) and strong opioids as a last resort in the absence of alternatives. In addition, psychotherapy, including cognitive behavioural therapy and mindfulness, is recommended as second-line treatment in combination with other therapies.

Pregabalin is also used in the treatment of epilepsy by blocking and modulating the α2 δ subunit of voltage-dependent calcium channels. There are studies showing that antiepileptics cause folate and vitamin B12 deficiency in epilepsy patients. In our study, we aimed to retrospectively analyse vitamin B12 and folic acid levels before and after treatment in patients using antiepileptics (anticonvulsants) for neuropathic pain.

DETAILED DESCRIPTION:
After the acceptance of the study (after obtaining ethics committee approval), patients who have been followed up for at least 6 months in the physical medicine and rehabilitation outpatient clinic with a diagnosis of neuropathic pain and who use pregabalin will be evaluated retrospectively (1-year records). Blood vitamin B12 and folate (folic acid) levels of the patients before and after pregabalin use will be determined. Patients will be evaluated whether there is a change in vitamin B12 and folic acid levels due to drug use.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90 years who have been diagnosed with neuropathic pain, whose vitamin B12 and folic acid levels have been analysed, who do not receive vitamin B12 and folic acid treatment, and who do not have diabetes mellitus, liver and kidney failure

Exclusion Criteria:

* Patients receiving vitamin B12 and folic acid therapy at the time of antiepileptic (anticonvulsant) drugs initiation, patients with hepatic and renal insufficiency

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were followed up for 6 months in the physical medicine and rehabilitation clinic with a diagnosis of neuropathic pain and who used antiepileptic (anticonvulsant) drugs will be retrospectively evaluated for the 6 months period (June-December 2024) before the ethics committee approval was obtained. Blood vitamin B12 and folate (folic acid) levels of the patients before and after antiepileptic drug use will be determined. Patients will be evaluated whether there is a change in vitamin B12 and folic acid levels depending on drug use.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Vitamin B12 level analysed before treatment (pre-treatment) (retrospective) | Within 1 month
  Vitamin B12 level (pg/mL) among the laboratory parameters analysed before antiepileptic treatment (pre-treatment) for neuropathic pain will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of neuropathic pain in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.
Vitamin B12 level analysed after treatment (post-treatment) (retrospective) | Within 1 month
  Vitamin B12 level (pg/mL) among the laboratory parameters analysed after antiepileptic treatment (post-treatment) for neuropathic pain will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of neuropathic pain in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.
Folic acid level analysed before treatment (pre-treatment) (retrospective) | Within 1 month
  Folic acid level (ng/mL), one of the laboratory parameters analysed before antiepileptic treatment for neuropathic pain (pre-treatment), will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of neuropathic pain in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.
Folic acid level analysed after treatment (post-treatment) (retrospective) | Within 1 month
  Folic acid level (ng/mL), one of the laboratory parameters analysed after antiepileptic treatment for neuropathic pain (post-treatment), will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of neuropathic pain in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.

SECONDARY OUTCOMES:
25-OH Vitamin D level analysed before treatment (pre-treatment) (retrospective) | Within 1 month
  D vitamini (25-OH Vitamin D) (ng/mL) among the laboratory parameters analysed before antiepileptic treatment (pre-treatment) for neuropathic pain will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of neuropathic pain in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.
25-OH Vitamin D level analysed after treatment (post-treatment) (retrospective) | Within 1 month
  25-OH Vitamin D (ng/mL) among the laboratory parameters analysed after antiepileptic treatment (post-treatment) for neuropathic pain will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of neuropathic pain in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

REFERENCES:
- [Background] Mula M, Sander JW. Negative effects of antiepileptic drugs on mood in patients with epilepsy. Drug Saf. 2007;30(7):555-67. doi: 10.2165/00002018-200730070-00001. PMID 17604407
- [Result] Aslan K, Bozdemir H, Unsal C, Guvenc B. The effect of antiepileptic drugs on vitamin B12 metabolism. Int J Lab Hematol. 2008 Feb;30(1):26-35. doi: 10.1111/j.1751-553X.2007.00910.x. PMID 18190464
- [Result] Linnebank M, Moskau S, Semmler A, Widman G, Stoffel-Wagner B, Weller M, Elger CE. Antiepileptic drugs interact with folate and vitamin B12 serum levels. Ann Neurol. 2011 Feb;69(2):352-9. doi: 10.1002/ana.22229. Epub 2011 Jan 19. PMID 21246600